CLINICAL TRIAL: NCT04020120
Title: Impact of Adult With Attention Deficit / Hyperactivity Disorder on Professional Activity, a Prospective Cohort Study
Brief Title: Assessment of the Professional Difficulties of Adult With Attention Deficit / Hyperactivity Disorder Patients
Acronym: WORKTDA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7482
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Attention Deficit Hyperactivity Disorder in Adults
Keywords: Prospective; Descriptive; Non-interventional; Monocentric
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADHD in professional activity: Adult ADHD patients in active employment at the time of inclusion or who were in employment within 3 months prior to inclusion
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — answer questionnaires

SUMMARY:
Attention Deficit/Hyperactivity Disorder (ADHD), which is common and well known in children, persists into adulthood in more than 60% of cases, with significant impact on quality of life. Professional domain is particularly impaired.

The investigators hypothesize that ADHD symptoms causes professional difficulties, on the emotional, cognitive, physical and relational levels.

The main objective of this study is to better characterize these professional difficulties at to follow-up these difficulties after one year. Difficulties will be assessed by questionnaires and semi-directive interview.

The secondary objective is to determine what factors modulate these difficulties and what compensation strategies are implemented to address the patients.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 18 to 62 years
* Diagnosis of attention deficit disorder with or without hyperactivity by a psychiatrist
* No treatment for ADHD in childhood or adolescence
* Patient who has been in a professional situation during the last 3 months

Exclusion criteria:

* Patient on sick leave or unemployed for more than 3 months
* Depressive episode in acute phase
* Subject with a mobility project that prevents follow-up for 1 year (planned move)
* Impossibility of providing the subject with informed information (subject in an emergency situation, difficulties in understanding the subject, mental retardation, illiteracy or insufficient command of the French language...)
* Subject under the protection of justice
* Subject under guardianship or curatorship

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who consulted at the psychiatric clinic of Strasbourg, aged 18 to 62, with a diagnosis of attention deficit disorder with or without hyperactivity assessed by a psychiatrist, and who have been in a working situation in the last 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The Work Limitations Questionnaire (WLQ-25) | 1 year
  It is a questionnaire with 25 items exploring 4 distinct dimensions: time management, physical demands, mental interpersonal demands and output demands.

SECONDARY OUTCOMES:
Maslach Burnout Inventory | 1 year
  It is a questionnaire with 22 items exploring 3 distinct dimensions: emotional exhaustion, deshumanization and personal achievement at work

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided